CLINICAL TRIAL: NCT05553002
Title: Does Improvement Towards a Normal Cervical Sagittal Configuration Aid in the Management of Lumbosacral Radiculopathy: A Randomized Controlled Trial
Brief Title: Does Improvement Towards a Normal Cervical Sagittal Configuration Aid in the Management of Lumbosacral Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Professor-chair of Physiotherapy Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cairo-11-2-15
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Cervical Lordosis Rehabilitation
Keywords: lumbosacral radiculopathy; Disc herniation; Cervical lordosis
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled study will be conducted at a research laboratory of our university. Participants will be randomly assigned to to either the treatment group or the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deneroll cervical extension traction (Experimental): The study group will receive 3-point bending cervical extension traction following the protocol of Deed Harrison . The duration of each session will start at approximately three minutes and increased one minute per session until reaching the goal of 20 minutes per session
  Interventions: Other: Deneroll cervical extension traction; Other: Traditional treatment
- Traditional treatment (Active Comparator): The participants will receive hot packs (15 minutes) and TENS therapy to control pain and eliminate the causal role of muscle spasms and/or tightness in changing the posture parameters.
  Interventions: Other: Traditional treatment

INTERVENTIONS:
Other: Deneroll cervical extension traction — Participants will lie flat on their back on the ground with their legs extended and arms by their sides. The denneroll will placed on the ground and positioned in the posterior aspect of the neck depending on the area to be addressed . The apex of the Denneroll orthotic will be placed in one of three regions based on lateral cervical radiographic displacements:
  1. In the upper cervical region (C2-C4) region.
  2. The apex of the Denneroll orthotic is placed in the mid-cervical region (C4-C6) region.
  3. The apex of the Denneroll orthotic is placed in the upper thoracic lower-cervical region (C6-T1) region.
  Arms: Deneroll cervical extension traction
Other: Traditional treatment — The participants will receive hot packs (15 minutes) and TENS therapy .During TENS application. Patients will be asked to adopt a prone position. The TENS therapy will be delivered at the lumbosacral region for 20 min. The frequency will set to 80 Hz and pulse width to 50 µs due to its analgesic effect . These conventional treatments will be repeated three times per week over the course of 10 weeks for 30 total sessions

SUMMARY:
A randomized controlled study with six months follow-up will be conducted to investigate the effects of sagittal head posture correction on 3D spinal posture parameters, back and leg pain, disability, and S1 nerve root function in patients with chronic discogenic lumbosacral radiculopathy . Participants will include 80 patients between 40 and 55 years experiencing chronic discogenic lumbosacral radiculopathy with a definite hypolordotic cervical spine and forward head posture and will be randomly assigned a comparative treatment control group and a study group. Both groups will receive TENS therapy and hot packs, additionally, the study group will receive the Denneroll cervical traction orthotic.

DETAILED DESCRIPTION:
Despite the fact that there is some evidence of a link between low back pain and head posture , there is limited experimental data to support a cause-and-effect relationship and interventional outcomes. Accordingly, a prospective, randomized, controlled study will be conducted at a research laboratory of our university to investigate if cervical curve restoration and forward head posture correction will have short and long term effects on three dimensional spinal posture parameters as well as lumbar radiculopathy management outcomes such as symptoms, disability, and neurophysiological findings .In this study we will use an orthotic cervical traction termed the Denneroll to help restore normal sagittal spinal configuration based on principles of 3-point bending traction methods. Interventions will be applied at a frequency of 3 times per week for 10 weeks and groups will be followed for an additional 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Absolute rotatory angle less than 25° and greater than 0.
* Anterior head translation distance greater than 15mm
* Confirmed chronic unilateral lumbosacral radiculopathy associated with L5-S1 lumbar disc prolapse .
* Symptoms lasting longer than 3 months

Exclusion Criteria:

* Previous history of lumbosacral surgery.
* Metabolic system disorder.
* Peripheral neuropathy.
* History of upper motor neuron lesion.
* Spinal canal stenosis.
* Rheumatoid arthritis.
* Osteoporosis

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-12-12 (Actual)

PRIMARY OUTCOMES:
The Change in cervical absolute rotatory angle | will be measured at three intervals :pretreatment, 10 weeks post treatment, and at six months of follow-up
  Cervical absolute rotatory angle is formed by two lines intersecting from the posterior body margins of C2-C7 and forward head distance
The Change in anterior head translation | will be measured at three intervals :pretreatment, 10 weeks post treatment, and at six months of follow-up
  anterior head translation is measured as the horizontal displacement of the posterior superior body corner of C2 vertebra relative to a vertical line extending superiorly from the posterior inferior body corner of C7..

SECONDARY OUTCOMES:
The change in 3D spinal posture parameters | will be measured at three intervals :pretreatment, 10 weeks post treatment, and at six months of follow-up
  Rasterstereography sagittal plane parameters (lumbar angles, thoracic angles, and trunk inclination), the frontal plane parameters (trunk imbalance and lateral deviation) and the transversal plane parameters (vertebral surface rotation and pelvis torsion) will be selected to cover the posture profile in three planes
The change in pain intensity | will be measured at three intervals :pretreatment, 10 weeks post treatment, and at six months of follow-up
  Measurement of pain will be performed by using a visual analogue scale (VAS). The subjects will be asked about the perception of pain using a 10-cm line with 0 (no pain) on one end and 10 (worst pain) on the other. subjects will be asked to place a mark along the line to denote their level of pain
The change in disability level | will be measured at three intervals :pretreatment, 10 weeks post treatment, and at six months of follow-up
  Disability will be measured using the Oswestry Disability Index. The total score is transferred onto a scale ranging from 0 to 100, where 0 indicates no disability and 100 indicates worst possible disability
The change in peak to peak amplitude of H reflex | will be measured at three intervals :pretreatment, 10 weeks post treatment, and at six months of follow-up
  The H-reflex (or Hoffmann's reflex) is a reaction of muscles after electrical stimulation of sensory fibers (Ia afferents stemming from muscle spindles) in their innervating nerves

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim M Moustafa, Professor, Principal Investigator — University of Sharjah
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No